CLINICAL TRIAL: NCT00057265
Title: A Randomized, Double Blind Trial of LdT (Telbivudine) Versus Lamivudine in Adults With Compensated Chronic Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV-02B-007
Record Dates: First submitted 2003-03-28; First posted 2003-03-31 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine; Lamivudine

INTERVENTIONS:
Drug: telbivudine or lamivudine

SUMMARY:
This study is being conducted to compare the safety and effectiveness of the investigational medication, LdT (Telbivudine) with Lamivudine, a drug currently approved by the US, European and Asian Health Authorities for the treatment of hepatitis B infection. The results for patients taking LdT will be compared to results for patients taking Lamivudine.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Hepatitis B, documented by Clinical history compatible with chronic HBV

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Patient is pregnant or breastfeeding
* Patient is co infected with hepatitis C virus (HCV), hepatitis D virus (HDV), HIV-1 or HIV-2.
* Patient previously received lamivudine or an investigational anti-HBV nucleoside or nucleotide analog at any time
* Patient has received interferon or other immunomodulatory treatment for HBV infection in the 12 months before screening for this study

Other protocol defined exclusion criteria may apply.

Ages: 16 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-02; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint: "therapeutic response", defined as reduction of serum HBV DNA to below 5 log10 copies/mL, coupled with normalization of serum alanine aminotransferase levels OR loss of detectable serum HBeAg.

SECONDARY OUTCOMES:
Secondary efficacy endpoints: Improvement of liver histology, serum HBV DNA changes, normalization of serum alanine aminotransferase levels, HBeAg and HBsAg loss and seroconversion.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (5):
  - Los Angeles, California
  - Orange, California
  - San Diego, California
  - Hackensack, New Jersey
  - Houston, Texas
- Seoul, South Korea
- Spain (2):
  - Barcelona
  - Valencia
- Bangkok, Thailand
- Istanbul, Turkey (Türkiye)
- London, United Kingdom

REFERENCES:
- [Derived] Zeuzem S, Gane E, Liaw YF, Lim SG, DiBisceglie A, Buti M, Chutaputti A, Rasenack J, Hou J, O'Brien C, Nguyen TT, Jia J, Poynard T, Belanger B, Bao W, Naoumov NV. Baseline characteristics and early on-treatment response predict the outcomes of 2 years of telbivudine treatment of chronic hepatitis B. J Hepatol. 2009 Jul;51(1):11-20. doi: 10.1016/j.jhep.2008.12.019. Epub 2009 Feb 12. PMID 19345439
- [Derived] Lai CL, Gane E, Liaw YF, Hsu CW, Thongsawat S, Wang Y, Chen Y, Heathcote EJ, Rasenack J, Bzowej N, Naoumov NV, Di Bisceglie AM, Zeuzem S, Moon YM, Goodman Z, Chao G, Constance BF, Brown NA; Globe Study Group. Telbivudine versus lamivudine in patients with chronic hepatitis B. N Engl J Med. 2007 Dec 20;357(25):2576-88. doi: 10.1056/NEJMoa066422. PMID 18094378